CLINICAL TRIAL: NCT06466980
Title: Study of Ventilator Associated Event During Intensive Care After Resuscitated Cardiac Arrest.
Acronym: VAE-ACR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0009
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest With Successful Resuscitation; Mechanical Ventilation
Keywords: Ventilator associated event; cardiac arrest; ventilator-acquired pneumonia; ventilator associated pneumonia
MeSH Terms: conditions — Heart Arrest; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ventilator associated event — Measure of incidence of Ventilator associated event

SUMMARY:
The aim is to describe the incidence, characteristics, risk factors and outcome of complications acquired under mechanical ventilation (called ventilator-associated events) according to the new CDC criteria, in a population of patients admitted in intensive care unit after cardiac arrest.

DETAILED DESCRIPTION:
Cardiac arrest (CA) survivors are frequently admitted to intensive care units. Despite improvements in management techniques, the prognosis of these patients remains poor, with mortality exceeding 90% for out-of-hospital CA and around 80% for in-hospital CA, along with a high risk of severe neurological issue.

The management of these patients in intensive care requires the use of invasive mechanical ventilation. Complications occurring under mechanical ventilation have been the subject of many researches. Early bacterial pneumonia or ventilator-acquired pneumonia appears as the primary cause of respiratory worsening, and several studies have already focused on their incidence and prevention. However, studies on the benefits of antibiotic therapy or antibiotic prophylaxis for early pulmonary infections are of tricky analysis, particularly when they do not consider respiratory condition or mortality for their primary outcome measure.

A new definition of complications associated with mechanical ventilation (VAEs) has been established by the Centers for Disease Control and Prevention (CDC) since 2013. It offers a more relevant tool for monitoring the impact of preventive measures on morbidity and mortality, with a more objective definition that goes beyond just tracking ventilator-associated pneumonia.

Several studies have since analyzed the incidence and impact of VAEs on cohorts of intensive care patients, confirming the association between VAEs and morbidity and mortality. However, to our knowledge, none have targeted a population of cardiac arrest survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Non-pregnant female
* Successfully resuscitated from cardiac arrest during primary care
* Invasive mechanical ventilation initiated during resuscitation and continued for at least 4 days
* No decision to limit life-sustaining therapies within 24 hours following admission to intensive care
* No requirement of arteriovenous circulatory support during intensive care management

Exclusion Criteria

- patients who opposed to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to intensive care unit after cardiac arrest at the South Francilien Hospital Center from January 2019 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number | at day 28
  Incidence of ventilator associated event

SECONDARY OUTCOMES:
Associated factors | at day 28
  Associated factors of ventilator associated event
number of pneumonias | at day 28
  Ventilator associated pneumonia according to the American Thoracic Society definition
time | at day 28
  Mechanical ventilation duration
number of deaths | at day 28
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Perbet S, Mongardon N, Dumas F, Bruel C, Lemiale V, Mourvillier B, Carli P, Varenne O, Mira JP, Wolff M, Cariou A. Early-onset pneumonia after cardiac arrest: characteristics, risk factors and influence on prognosis. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1048-54. doi: 10.1164/rccm.201102-0331OC. PMID 21816940